CLINICAL TRIAL: NCT05167409
Title: A Phase II Study (With Safety run-in) of Evorpacept (ALX148) in Combination With Cetuximab and Pembrolizumab in Patients With Refractory Microsatellite Stable Metastatic Colorectal Cancer
Brief Title: A Study of Evorpacept (ALX148) With Cetuximab and Pembrolizumab for Refractory Microsatellite Stable Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: ALX Oncology Inc. (Industry); Merck Sharp & Dohme LLC (Industry); Eli Lilly and Company (Industry); Criterium, Inc. (Industry); Academic GI Cancer Consortium (AGICC) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0110.cc; NCI-2022-02019 (Other Grant/Funding Number: CTRP); AGICC-ALX148 21CRC01 (Other: AGICC)
Record Dates: First submitted 2021-09-27; First posted 2021-12-22 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Microsatellite Stable Metastatic Colorectal Cancer
Keywords: evorpacept (ALX148); Cetuximab; Pembrolizumab; CRC; colorectal cancer; microsatellite stable; MSS; CD47; SIRPa
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ALX148; Cetuximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Evorpacept (ALX148) + cetuximab + pembrolizumab (Experimental): Evorpacept (ALX148) + cetuximab + pembrolizumab. Evorpacept (ALX148) 15 mg/kg IV weekly, cetuximab 400 mg/m2 once then 250 mg/m2 weekly, and pembrolizumab 200 mg every 3 weeks
  Interventions: Drug: Evorpacept (ALX148); Drug: Cetuximab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Evorpacept (ALX148) — IV QW
  Other Names: evorpacept
Drug: Cetuximab — IV QW
  Other Names: Erbitux
Drug: Pembrolizumab — IV Q3W
  Other Names: Keytruda

SUMMARY:
This Phase 2 clinical study will evaluate evorpacept (ALX148) in combination with cetuximab and pembrolizumab for refractory microsatellite stable metastatic colorectal cancer

DETAILED DESCRIPTION:
This is an open-label, multi-center, single-arm phase II clinical trial (with safety run-in) evaluating the combination of evorpacept (ALX148), cetuximab, and pembrolizumab in patients with metastatic microsatellite stable colorectal cancer who have progressed on at least 2 lines of systemic therapy. A subset of patients will undergo study-related biopsies. There will be a safety run-in stage followed by a dose expansion stage. Patients in both stages will continue to receive study therapy until disease progression according to RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Have a diagnosis of metastatic colorectal cancer previously treated with at least two lines of therapy for unresectable/metastatic disease
* Have microsatellite stable disease
* Adequate hematologic and end organ function

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patients with known MSI-high status or known mismatch repair deficiency (dMMR)
* Patients in whom both mismatch repair and microsatellite stability status are unknown
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to any of the study medications or their classes
* Left-sided (at or distal to the splenic flexure) RAS/BRAF wild-type metastatic colorectal cancer who are EGFR inhibitor naïve.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti PD L2, anti-CD47, or anti-SIRPα agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Recommended dose (RD) of evorpacept (ALX148) in combination with cetuximab and pembrolizumab 1.(mg/kg) | 4 months
  To determine the recommended dose (RD) of evorpacept (ALX148) in combination with cetuximab and pembrolizumab
Objective response rate (ORR, per RECIST v1.1) (%) | 6 months
  To determine the objective response rate (ORR), defined as partial response or complete response, with evorpacept (ALX148), cetuximab, and pembrolizumab using RECIST v1.1 in patients with microsatellite stable (MSS) metastatic colorectal cancer (mCRC) who have progressed on at least two lines of standard therapy

SECONDARY OUTCOMES:
Disease control rate per RECIST v1.1. (%) | 24 months
  To determine the disease-control rate (DCR), defined as stable disease, partial response, or complete response with evorpacept (ALX148), cetuximab, and pembrolizumab using RECIST v1.1
Duration of response per RECIST v1.1. (months) | 24 months
  To determine the duration of response (DOR) with evorpacept (ALX148), cetuximab, and pembrolizumab, defined as the time from response (partial or complete) to progression
Progression-free survival (PFS, per RECIST v1.1) (months) | 48 months
  To determine the progression-free survival (PFS) with evorpacept (ALX148), cetuximab, and pembrolizumab, defined as the time from enrollment to the first observation of progression using RECIST v1.1 or death from any cause
Overall survival (OS) | 48 months
  To determine the overall survival (OS) with evorpacept (ALX148), cetuximab, and pembrolizumab, defined as the time from enrollment to death from any cause
First cycle dose-limiting toxicities in the safety run-in stage | 4 months
  To determine the first cycle dose-limiting toxicities (DLT) of evorpacept (ALX148), cetuximab, and pembrolizumab in stage 1
Safety and tolerability according to the NCI CTCAE v5.0 | 48 months
  To evaluate the safety and tolerability of evorpacept (ALX148), cetuximab, and pembrolizumab, defined and graded according to the NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lentz, MD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rutgers Cancer insititute, New Brunswick, New Jersey
  - Inova Schar Cancer Institute, Fairfax, Virginia